CLINICAL TRIAL: NCT04907877
Title: Role of Nutritional Support With Probiotics in Adult Outpatients With Symptomatic COVID-19: a Randomized Dietary Study
Brief Title: Bifido- and Lactobacilli in Symptomatic Adult COVID-19 Outpatients
Acronym: ProCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Biotic Sp. z o.o. (Industry)
Responsible Party: Principal Investigator, Sergei Gerasymov, MD, PhD, Principal Investigator, Nordic Biotic Sp. z o.o.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-Resp-CoV-2-A0003
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): NordBiotic ImmunoVir, a mixute of bidido- and lactobacteria administered in a dose of 5 billion once a day for 28 days
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Maltodextrine administered once a day for 28 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic will be taken 1 time a day before breakfast for 28 days.
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo will be taken 1 time a day before breakfast for 28 days.
  Arms: Placebo

SUMMARY:
There is evidence that some types of probiotics play a role in alleviation of symptoms of acute respiratory tract infections and bursting immune response to respiratory and enteric viruses. Available data serves a rationale for the study exploring a role of nutritional support with probiotics in adult outpatients with COVID-19. Hypothesis of the study is that a proposed mixture of lactobacilli and bifidobacteria facilitate faster recovery from COVID-19 and enhance specific immune response to SARS-CoV-2 antigens.

DETAILED DESCRIPTION:
One hundred adults with confirmed (PCR or antigen test) symptomatic COVID-19 lasting upto 5 days will be screened for the study. When the subject meets enrollment criteria, he/she will be randomized to take an investigational product (probiotic, test dietary supplement, TDS), a mixture of lactobacilli and bifidobacteria or placebo 1 time a day before breakfast for 28 days after enrollment. During observation, the patient will keep Respiratory Illness Diary. Blood serum will be collected at baseline, day 0-5 (Nurse Visit 1), after 28-35 days (Nurse visit 2), and 6 months (Nurse visit 3) for evaluation of anti-SARS-CoV-2 antibodies to nucleocapsid and spike antigents. In 3 months, investigator/family physician will collect Post-COVID-19 Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 - ≤ 65 years;
2. Male or non-pregnant female;
3. Informed virtual pre-consent and paper signed consent forms;
4. Confirmed symptomatic COVID-19 lasting 0-5 days;
5. Subject understands and agrees to comply with study procedures including triple blood analysis for anti-SARS-CoV-2 IgG;

Exclusion Criteria:

1. Risk for the complicated course of COVID-19 due to:

   1.1. Hypertension; 1.2. Diabetes mellitus; 1.3. Immunosuppressive conditions; 1.4. Chronic pathology of the respiratory system ; 1.5. Chronic pathology of the cardiovascular system ; 1.6. Malignant tumor ; 1.7. Systemic inflammatory connective tissue disease ; 1.8. Cerebrovascular disease ; 1.9. Chronic hepatitis. Hepatic cirrhosis; 1.10. Inflammatory bowel diseases ; 1.11. Chronic kidney disease ;
2. Drug or alcohol abuse as suspected by investigator;
3. History of persistent diarrhea of any cause;
4. Use of pre- or probiotics during the last 2 weeks before enrollment;
5. Allergy to any components of the TDS;
6. Technical difficulties to perform virtual study visits.
7. Inability to perform a blood test for antibodies after 6 months
8. Inability to swallow capsules, or choking / coughing while eating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Global symptom score | 10 days
  Clinical score of Coronavirus disease-19; minimal score 0 (healthy), maximal score 36 (worst disease)

SECONDARY OUTCOMES:
8 - point ordinal severity scale of coronavirus disease-19 | 28 days
  World Health Organization scale; score 0 - healthy, score 8 - death
Time to recovery | 28 days
  Day when patient symptom score is 0
Percent of completely recovered patients | 28 days
  Patients with symptom score is 0
Hospitalization rate | 28 days
  Percent hospitalized due to COVID-19

OTHER OUTCOMES:
Anti-SARS-CoV-2 antibodies IgG response | Days 0-5, day 28-35, month 6th
  Antibody titer to NCP and spike antigen

CONTACTS AND LOCATIONS:
Overall Officials: Zoriana Hoda, MD, Study Director — Lviv State Laboratory Center, Ministry of Health of Ukraine
Locations (3):
- Ukraine (3):
  - Hemo Medica Ukraine Ltd, Uzhhorod, Zakarpatska
  - Lviv State Center for Disease Control and Prevention, Lviv
  - 3rd City Clinical Hospital of Lviv, Lviv

IPD SHARING:
Plan to Share IPD: No
Not applicable as not decided yet

REFERENCES:
- [Result] Pan L, Mu M, Yang P, Sun Y, Wang R, Yan J, Li P, Hu B, Wang J, Hu C, Jin Y, Niu X, Ping R, Du Y, Li T, Xu G, Hu Q, Tu L. Clinical Characteristics of COVID-19 Patients With Digestive Symptoms in Hubei, China: A Descriptive, Cross-Sectional, Multicenter Study. Am J Gastroenterol. 2020 May;115(5):766-773. doi: 10.14309/ajg.0000000000000620. PMID 32287140
- [Result] Smyk W, Janik MK, Portincasa P, Milkiewicz P, Lammert F, Krawczyk M. COVID-19: Focus on the lungs but do not forget the gastrointestinal tract. Eur J Clin Invest. 2020 Sep;50(9):e13276. doi: 10.1111/eci.13276. Epub 2020 Jul 5. PMID 32406522
- [Result] Westermann C, Gleinser M, Corr SC, Riedel CU. A Critical Evaluation of Bifidobacterial Adhesion to the Host Tissue. Front Microbiol. 2016 Aug 5;7:1220. doi: 10.3389/fmicb.2016.01220. eCollection 2016. PMID 27547201
- [Result] Van Tassell ML, Miller MJ. Lactobacillus adhesion to mucus. Nutrients. 2011 May;3(5):613-36. doi: 10.3390/nu3050613. Epub 2011 May 20. PMID 22254114
- [Result] Olaimat AN, Aolymat I, Al-Holy M, Ayyash M, Abu Ghoush M, Al-Nabulsi AA, Osaili T, Apostolopoulos V, Liu SQ, Shah NP. The potential application of probiotics and prebiotics for the prevention and treatment of COVID-19. NPJ Sci Food. 2020 Oct 5;4:17. doi: 10.1038/s41538-020-00078-9. eCollection 2020. PMID 33083549
- [Result] Yeoh YK, Zuo T, Lui GC, Zhang F, Liu Q, Li AY, Chung AC, Cheung CP, Tso EY, Fung KS, Chan V, Ling L, Joynt G, Hui DS, Chow KM, Ng SSS, Li TC, Ng RW, Yip TC, Wong GL, Chan FK, Wong CK, Chan PK, Ng SC. Gut microbiota composition reflects disease severity and dysfunctional immune responses in patients with COVID-19. Gut. 2021 Apr;70(4):698-706. doi: 10.1136/gutjnl-2020-323020. Epub 2021 Jan 11. PMID 33431578
- [Result] Chai W, Burwinkel M, Wang Z, Palissa C, Esch B, Twardziok S, Rieger J, Wrede P, Schmidt MF. Antiviral effects of a probiotic Enterococcus faecium strain against transmissible gastroenteritis coronavirus. Arch Virol. 2013 Apr;158(4):799-807. doi: 10.1007/s00705-012-1543-0. Epub 2012 Nov 28. PMID 23188495
- [Result] Miettinen M, Pietila TE, Kekkonen RA, Kankainen M, Latvala S, Pirhonen J, Osterlund P, Korpela R, Julkunen I. Nonpathogenic Lactobacillus rhamnosus activates the inflammasome and antiviral responses in human macrophages. Gut Microbes. 2012 Nov-Dec;3(6):510-22. doi: 10.4161/gmic.21736. Epub 2012 Aug 16. PMID 22895087
- [Result] Nakayama Y, Moriya T, Sakai F, Ikeda N, Shiozaki T, Hosoya T, Nakagawa H, Miyazaki T. Oral administration of Lactobacillus gasseri SBT2055 is effective for preventing influenza in mice. Sci Rep. 2014 Apr 10;4:4638. doi: 10.1038/srep04638. PMID 24717726
- [Result] Gao X, Huang L, Zhu L, Mou C, Hou Q, Yu Q. Inhibition of H9N2 Virus Invasion into Dendritic Cells by the S-Layer Protein from L. acidophilus ATCC 4356. Front Cell Infect Microbiol. 2016 Oct 25;6:137. doi: 10.3389/fcimb.2016.00137. eCollection 2016. PMID 27826541
- [Result] Vouloumanou EK, Makris GC, Karageorgopoulos DE, Falagas ME. Probiotics for the prevention of respiratory tract infections: a systematic review. Int J Antimicrob Agents. 2009 Sep;34(3):197.e1-10. doi: 10.1016/j.ijantimicag.2008.11.005. Epub 2009 Jan 28. PMID 19179052
- [Result] Zimmermann P, Curtis N. The influence of probiotics on vaccine responses - A systematic review. Vaccine. 2018 Jan 4;36(2):207-213. doi: 10.1016/j.vaccine.2017.08.069. Epub 2017 Sep 18. PMID 28923425
- [Derived] Kolesnyk PO, Paliy IH, Sydorchuk LP, Hoda ZP, Ivanchenko NO, Lych OS, Huley NR, Matsyura OI, Slyuzar ZL, Gerasymov SV. The role of nutritional support with probiotics in outpatients with symptomatic acute respiratory tract infections: a multicenter, randomized, double-blind, placebo-controlled dietary study. BMC Nutr. 2024 Jan 4;10(1):4. doi: 10.1186/s40795-023-00816-8. PMID 38178223